CLINICAL TRIAL: NCT06686368
Title: Comparative Efficacy of I-DROP®MGD Versus Competing Eye Drops in Managing Evaporative Dry Eye: A Pilot Randomized Controlled Trial
Brief Title: Comparative Efficacy Study to Demonstrate the Non-inferiority of I-DROP® MGD Versus 2 Competitor Eye Drops in Managing Evaporative Dry Eye
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: I-MED Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR001-2024
Record Dates: First submitted 2024-10-23; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Evaporative Dry Eye Disease
Keywords: Dry Eye Disease; Lubricant eye drops; Meibomian Gland Dysfunction; Evaporative dry eye
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: in vivo, human patient with confirmed Evaporative dry eye disease
Who Masked: Participant, Care Provider, Investigator
Masking Description: All products will have their label removed and placed a white sticker showing the group (A or B or C). Products with be put in a white box with the letter indicated on it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- I-DROP MGD (Experimental): High Molecular weight hyaluronic acid + PC containing lubricant eye drop Receiving lubricant eye drops with high molecular weight hyaluronic acid
  Interventions: Device: I-DROP MGD
- Thealoz Duo (Active Comparator): Low Molecular weight hyaluronic acid + Trehalose containing lubricant eye dropReceiving lubricant eye drops with low molecular weight hyaluronic acid
  Interventions: Device: Theloze Duo
- Systane Complet PF (Active Comparator): No hyaluronic acid containing lubricant eye drop Receiving lubricant eye drops without hyaluronic acid
  Interventions: Device: Systane Complete PF

INTERVENTIONS:
Device: I-DROP MGD — All drops are to be used for 28-30 days, twice daily with assessment done at Day 0, 30 minutes post-installation at day 0, day 7 and day 28/30
  Arms: I-DROP MGD
Device: Theloze Duo — All drops are to be used for 28-30 days, twice daily with assessment done at Day 0, 30 minutes post-installation at day 0, day 7 and day 28/30
  Arms: Thealoz Duo
Device: Systane Complete PF — All drops are to be used for 28-30 days, twice daily with assessment done at Day 0, 30 minutes post-installation at day 0, day 7 and day 28/30
  Arms: Systane Complet PF

SUMMARY:
A Pilot Comparative study between I-DROP MGD vs two commercially available lubricant eye drops for the management of evaporative dry eye

DETAILED DESCRIPTION:
Pilot, randomized, double-blind, prospective, non-inferiority study to demonstrate the safety and efficacy of I-DROP MGD vs two commercially available preservative-free lubricant eye drops for the management of evaporative dry eye

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and signed an information consent form.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Has dry eye disease as per the TFOS DEWS II definition with a clear moderate to severe evaporative Dry Eye:

  * OSDI ≥ 13
  * And TBUT < 10 seconds
  * And >5 spots of corneal fluorescein staining OR > 9 conjunctival spots
  * Meibomian Gland score of 1 or higher using NEI grading criteria.

Exclusion Criteria:

* Is participating in any concurrent clinical or research study.
* Is wears contact lenses.
* Is using any systemic medications that could impact the aqueous tear layer, including antihistamines, vitamin A analogues, phenothiazines, anti-anxiety drugs, antidepressants, and other medications with anticholinergic activity.
* Has undergone eye surgery involving the cornea or conjunctiva.
* Aqueous deficient DED patients.
* Is currently or has used any of the study drops in the last 3 months.
* Has any known allergy or intolerance to any of the study drops.
* Has any known active ocular disease such as allergies and/or infection or any ocular disease that in the opinion of the investigator may affect a study outcome variable
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable (e.g. uncontrolled autoimmune disease or uncontrolled immunodeficiency disease).
* Has known sensitivity to sodium fluorescein.
* Is pregnant, lactating or planning a pregnancy at the time of enrolment?
* Unwilling to stop using their habitual artificial tears for the study.
* Has been fitted with punctal plugs within 30 days before the study screening visit.
* Contact lens users can still qualify for the study, however, participants should restrain their contact lens use to a very minimum during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Fluorescein Tear Break-Up Time (FTBUT) in seconds | Day 1 - 30 minutes post installation
  The primary outcome of the study is FBUT at 30 minutes post-installation

SECONDARY OUTCOMES:
Fluorescein Tear Break-Up Time (FTBUT) in seconds | Day 7 - day 28
  One of the secondary endpoints is FTBUT at day 7 and day 28
Tear Meniscus Height (TMH) in milimiters | Day 1 - Day 7 - day 28
  One of the secondary endpoints is TMH at day 1 (30 minutes post-installation), 7 and day 28
Osmolarity in mOsm/L | Day 1 - Day 7 - day 28
  One of the secondary endpoints is osmolarity at day 1 (30 minutes post-installation), 7 and day 28
Number of Corneal and Conjunctival spots | Day 7 - day 28
  One of the secondary endpoints is Corneal and conjunctival spots at day 7 and day 28
Ocular Surface and Disease Index (OSDI) score | Day 7 - day 28
  One of the secondary endpoints is OSDI score at day 7 and day 28

IPD SHARING:
Plan to Share IPD: No